CLINICAL TRIAL: NCT05025176
Title: Hypotension Prediction Index: Correlations Between Invasive and Non-invasive Pressure Points
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 1791102
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery requiring Invasive arterial pressure monitoring: Patients undergoing elective surgery that requires Invasive arterial pressure monitoring as standard of care.
  Interventions: Device: Non invasive arterial pressure monitoring

INTERVENTIONS:
Device: Non invasive arterial pressure monitoring — Non invasive arterial pressure monitoring

SUMMARY:
To evaluate the clinical performance of the Hypotension Prediction Index obtained from the continuous, non-invasive Clear Sight monitor.

DETAILED DESCRIPTION:
To evaluate the clinical performance of the Hypotension Prediction Index obtained from the continuous, non-invasive ClearSight monitor.

ELIGIBILITY:
Inclusion Criteria:

* All Patients 18 years or older undergoing surgery with the use of general anesthesia and with planned arterial catheter placement and use of the HPI monitor.

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults ( infants, children teenagers)
* Pregnant Women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patents undergoing surgery with a planner arterial catheter placement
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
HPI | During surgical procedure
  Hypotension Prediction Index obtained from continuous, non-invasive ClearSight monitor will not differ significantly from the HPI concurrently obtained from the standard of care invasive radial arterial pressure monitor

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Health System, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarhadi K, Hamman J, Avila J, Jian Z, Fleming NW. Hypotension prediction index: comparison between invasive and non-invasive pressure inputs. BMC Anesthesiol. 2025 Apr 29;25(1):221. doi: 10.1186/s12871-025-03086-y. PMID 40301710